CLINICAL TRIAL: NCT03414151
Title: Gut Microbiome and Metabolic Dysfunction in Antipsychotic Naïve Patients
Brief Title: Gut Microbiome in AP Naive
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Margaret Hahn, Clinician/Scientist, Centre for Addiction and Mental Health
Other Study IDs: 030/2017
Record Dates: First submitted 2017-10-28; First posted 2018-01-29 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Psychotic Disorder; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood serum; fecal sample (collected in OMNIgene•GUT, DNA Genotek Ottawa, ON)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational - Case Arm: All participants will be placed in this arm or group if they have an eligible psychiatric diagnosis as a case (there is no randomization procedure)
  Interventions: Other: Observation
- Observational - Healthy Control Arm: All participants will be placed in this arm if they are healthy controls (there is no randomization procedure)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention administered.

SUMMARY:
Antipsychotic (AP) medications are currently the cornerstone of treatment for schizophrenia (SCZ), with off-label prescription rapidly increasing in youth, with an established two-fold increase in standardized mortality ratio attributable to cardiovascular disease in this population. However, APs have been associated with common and serious metabolic adverse effects including weight gain and diabetes, to which youth are disproportionally vulnerable. The Gut Microbiome (GMB) has been suggested as a potential target warranting further study as a mechanism of AP induced weight gain and has also been linked directly with cognition and behavior. It is hypothesized that there will be changes in the gut microbiome overtime with treatment correlated with metabolic measures and that APs will produce changes in glucose tolerance, insulin sensitivity, adipokines, glucagon like peptide (GLP)-1, lipids, fasting glucose, body weight, and cognition.

DETAILED DESCRIPTION:
The objectives of the study are to examine the gut microbiome composition and diversity in patients with schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum and other psychotic disorder at 6 weeks and 3 months post antipsychotic initiation. Furthermore, the team aims to investigate causality of antipsychotic (AP)-induced changes in the GMB in relation to metabolic changes. This will be accomplished by transplanting human gut microbiota from patients initiating an AP treatment into germ-free mice (independent animal protocol). The final objective is to observe changes in cognition associated with changes in metabolic factors and gut microbiome.

The hypotheses of the study are twofold: the primary hypothesis is that there will be changes in the gut microbiome overtime with treatment correlated with metabolic measures (i.e. weight, insulin sensitivity, glucose tolerance, lipids) due to treatment in antipsychotic naïve patients, and the gut microbiome of treated patients transplanted into germ-free mice will induce similar metabolic proving causality (separate animal protocol). The secondary hypothesis is that APs will produce changes psychopathology and cognitive outcome measures which will correlate with changes in gutmicrobiome.

Participants will include individuals who are either antipsychotic naïve or have not taken antipsychotics for at least 3 months prior to study participation. Participants will be between 12 and 35 years of age with a diagnosis of schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum and other psychotic disorder, as per DSM-V criteria. Participants will be enrolled to reach n=25 complete data sets. Participants who drop out or who are withdrawn will be replaced.

Following provision of written informed consent, participants will be assessed for suitability for inclusion in the study based on the inclusion and exclusion criteria. Participants will be seen across 5 timepoints, including a screening and baseline visit, as well as 3 follow-up appointments.

Within-group analyses will be conducted to evaluate changes in participants at different time points on measures including anthropometric measures, clinical scales, and fasting bloodwork results. Microbiome analysis will include α-diversity metrics for each sample and β-diversity measures (weighted and unweighted unifrac, Specifically we will analyze changes in the microbiome pre- and post- antipsychotic treatment and whether changes in the microbiome associate with other clinical and biochemical measures. We will also determine whether patients that develop metabolic side effects with antipsychotic treatment have different microbial profiles than those who do not develop these side effects.

Whole body insulin sensitivity is calculated based on the original description by Matsuda at baseline and endpoint. HOMA-IR will be calculated at baseline, week 6, and week 12 to determine change in insulin resistance over time.

A blood sample will be collected for DNA extraction to examine for the genes that that are hypothesized to be associated to response or side effects following antipsychotic medication. Fecal DNA analyses will be completed at McMaster University. Stool samples will be collected from participants at baseline, weeks 3 and 6. Participants will be given stool collection kits (OMNIgene•GUT, DNA Genotek Ottawa, ON). Participants will return the sample at their earliest convenience. Once returned, samples will be immediately frozen and stored at -80°C.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-35
* Antipsychotic naïve or antipsychotic treatment for equal to or less than 2 weeks within the past 3 months; the minimum AP dose will be left to the discretion of the PI
* DSM-5 diagnosis (using SCID-IV-TR with supplemental questions from SCID-5 or SCID-5) of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, and brief psychotic disorder, psychotic disorder NOS. and/or antipsychotic treatment for schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum and other psychotic disorder.

Exclusion Criteria:

* Previous antipsychotic treatment (greater than two weeks within the preceding 3 months)
* Presence of DSM-5 diagnosis which is not schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum and other psychotic disorder
* Use of any other medications for treatment of lipids, glucose, or weight as deemed to be clinically significant by the PI
* Use of other medications where the dose has changed within the past 6 weeks which are deemed by the PI to be clinically significant
* Pregnancy
* Eating disorder - active or previous
* Major medical or surgical event within the preceding 3 months
* Acute suicidal risk
* Irritable bowel disease, Crohn's disease, and/or diverticulitis/diverticulosis
* Type I diabetes, kidney/liver disease, and/or cancer
* Organ transplant
* Moderate to severe alcohol use , use of street drugs, and/or cannabis use (as deemed by PI)
* Immunosuppressants and/or anti-inflammatory medications
* Antibiotic/probiotic use within past 4 weeks
* Any other medical conditions or lifestyle habits deemed by the PI to impact the integrity of the sample/microbiota

Ages: 12 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants will include individuals who are either antipsychotic naïve or have not taken antipsychotics for at least 3 months prior to study participation. Participants will be between 12 and 35 years of age with a diagnosis of schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum and other psychotic disorder, as per DSM-V criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in Gut microbiome and DNA | 12 weeks (baseline, week 6, week 12)
  Patients will collect fecal samples at home using our well-established protocol at baseline, 6 weeks, and 12 weeks. Participants will be provided a kit containing a sterile specimen container and a cooling pad, as well as a stool collection tube for DNA analyses (OMNIgene•GUT, DNA Genotek Ottawa, ON). Patients will be instructed to transfer several grams of the feces into the specimen container and place the sample in the 2 bioharzard bags and then store in the freezer. On the day of their appointment they will transport the sample on the cooling pad (previously placed in the freezer) to their appointment. When the patient delivers the sample to the research staff, it will be immediately placed in a -80ºC freezer prior to being analyzed. These analyses with fecal samples will be conducted at McMaster University at the Farncombe Family Institute.

SECONDARY OUTCOMES:
Oral glucose tolerance test | 12 weeks (baseline and week 12)
  Following collection of baseline samples, a standard glucose drink (75mg) is given orally, and a blood sample of insulin and glucose is obtained exactly 1 hour and 2 hours after the standard glucose drink is administered. Blood will be drawn at a total of 4 time points. Serums which will be collected during this procedure include fasting glucose; fasting insulin; leptin, fasting free fatty-acids, c-peptide, cortisol; Glucagon-like polypeptide-1 (GLP-1), glucagon inhibitory peptide (GIP),cytokines, ghrelin related to weight gain and glucose metabolism.
Height | 12 weeks
  Height (cm) will be collected at the initial study visit
Weight | 12 weeks
  Weight (kg) will be collected at each study visit
Blood pressure | 12 weeks
  Blood pressure will be measured at each study visit (sys/dia)
Heart Rate | 12 weeks
  Heart rate will be measured at each study visit (BPM)
Waist Circumference | 12 weeks
  Waist circumference (cm) will be measured at each study visit
BMI | 12 weeks
  BMI (kg/m^2) will be calculated at each study visit
Prolactin | 12 weeks (baseline, week 6, week 12)
  Prolactin levels will be collected via blood work.
Liver enzymes | 12 weeks (baseline, week 6, week 12)
  Liver enzymes including ALT (unit/L), ALP (unit/L), and AST (unit/L) will be collected via bloodwork.
Bilirubin | 12 weeks (baseline, week 6, week 12)
  Bilirubin (mcmol/L) values will be collected via bloodwork.
GGT | 12 weeks (baseline, week 6, week 12)
  GGT (unit/L) values will be collected via bloodwork.
Albumin | 12 weeks (baseline, week 6, week 12)
  Albumin (g/L) values will be collected via bloodwork.
HbA1c | 12 weeks (baseline, week 6, week 12)
  HbA1c will be collected via bloodwork.
Fasting blood work | 12 weeks (baseline, week 6, week 12)
  Fasting bloodwork values including lipids (mmol/L), glucose (mmol/L), AAP serum levels (mmol/L), and electrolytes (mmol/L) will be collected via bloodwork.
CBC | 12 weeks (baseline, week 6, week 12)
  CBC values will be collected via blood work.
Thyroid Stimulating Hormone (TSH) | 12 weeks (baseline, week 6, week 12)
  TSH (mIU/L) values will be collected via blood work.
Insulin | 12 weeks (baseline, week 6, week 12)
  Insulin (pmol/L) values will be collected via blood work.
Leptin | 12 weeks (baseline, week 6, week 12)
  Leptin values will be collected via blood work.
Free Fatty Acids (FFA) | 12 weeks (baseline, week 6, week 12)
  FFA values will be collected via blood work.
C-peptide | 12 weeks (baseline, week 6, week 12)
  C-peptide (ng/mL) values will be collected via blood work.
Cortisol | 12 weeks (baseline, week 6, week 12)
  Cortisol (mcg/dL) values will be collected via blood work.
DNA | Baseline measure
  DNA will be collected via blood work.
Brief Psychiatric Rating Scale 18 item (BPRS) | 12 weeks (baseline, week 6, week 12)
  The BPRS is a rater administered interview evaluating psychiatric symptoms. Total scores range between 18 and 126, with higher scores indicating greater severity of symptoms. Total scores are calculated by adding all individual item scores.
The Positive and Negative Symptom Questionnaire (SANS) | 12 weeks (baseline, week 6, week 12)
  The SANS is a rater administered interview evaluating positive and negative symptoms in psychosis. Total scores range from 0 to 110, with higher scores indicating greater severity of symptoms.Total scores are calculated by adding all individual item scores.
Clinical Global Impression (CGI) | 12 weeks (baseline, week 6, week 12)
  The CGI is a rater-observed measure which evaluates overall mental illness severity. The score ranges from 1 to 7, with a higher score indicating greater severity of symptoms.
The Calgary Depression Scale for Schizophrenia (CDSS) | 12 weeks (baseline, week 6, week 12)
  The CDSS is a rater administered interview evaluating the presence and severity of depressive symptoms in schizophrenia. The total score ranges from 0 to 27, with higher scores indicating a greater severity. Total scores are calculated by adding all individual item scores.
Quality of Life Scale (QLS) | 12 weeks (baseline, week 6, week 12)
  The QLS is a questionnaire measuring the functioning of outpatient schizophrenia patients and measures the quality of relationships, occupational roles, and personal experiences. Subscale scores include Interpersonal Relations (range 0-72), Instrumental Role (range 0-36), Intrapsychic Function (range 0-63), Common Objects and Activities (range 0-18). The total score is then calculated by adding all the individual items together for a total score range of between 0-189. Higher scores across all variables indicate poorer quality of life. Total scores are calculated by adding all individual item scores.
Birchwood Social Functioning Scale (BSFS) | 12 weeks (baseline, week 6, week 12)
  The BSFS is a scale used to measure quality of social functioning. Subscales include Social Engagement/Withdrawal (range 0-15), Interpersonal Communication (range 0-9), Independence-Performance (range 0-39), Recreation (range 0-45), Prosocial (range 0-66), Independence-Competence (range 0-39), and Occupation/Employment (range 0-10). Higher scores indicate better social functioning. Scores are calculated by adding all individual item scores.
UKU Side Effects Scale | 12 weeks (all time points)
  A rater-administered evaluation of side-effects related to psychopharmacological drugs. Ratings are given on a scale of 0-3, with higher scores indicating greater severity. An overall score, assigned by rater impression, is given to indicate overall incapacity due to side-effects.
Abnormal Involuntary Movement Scale (AIMS) | 12 weeks (baseline, week 12)
  A rater-administered evaluation of tardive dyskinesia. Scores are assigned across 3 categories including facial and oral movement, extremity movement, and trunk movement. There are no subscale scores however a global rating is given from a range of 0-4 based on the average of the categorical ratings, with higher scores indicated greater severity.
Barnes Akathisia Scale (BAS) | 12 weeks (baseline, week 12)
  A rater-administered evaluation of akathisia. A rating of 0-3 is given for objective and subjective awareness of fidgeting, respectively, as well as for distress related to movement. A global score, as calculated on the average of all individual scores, is assigned on a scale of 0-5.
Simpson Angus Scale (SAS) | 12 weeks (baseline, week 12)
  A rater-administered evaluation of extrapyramidal symptoms. Scores range from normal (score 0-3), minimal degree of movement disorder (score 3-5), clinically significant degree of movement disorder (score 6-11), and severe degree of movement disorder (score 12-17). Items are rated individually (i.e. no composite score).
Food Cravings Questionnaire (FCQ) | 12 weeks (baseline, week 6, week 12)
  A self-administered rating of food cravings and eating behaviours, both trait and state. A total score is calculated by adding all scores together. Higher scores indicate heightened trait and or state behaviour.
Visual Analog Scale (VAS) | 12 weeks (baseline, week 6, week 12)
  A self-administered rating of food cravings where participants mark on a continuum . The location of the mark is then measured (cm) for each item. Some items are reverse scored so individual items need to be reviewed for context. Only individual item scores are assigned (i.e. no total score assigned).
Harvard Youth/Adolescent Questionnaire (YAQ) | 12 weeks (baseline, week 6, week 12)
  A self-administered food frequency questionnaire designed for older children and adolescents. Individuals scores are evaluated for nutritional breakdown. This is a qualitative self-report assessment.
International Physical Activity Questionnaire (IPAQ) | 12 weeks (baseline and week 12)
  A rater administered questionnaire evaluating health-related physical activity. A composite score is calculated by combining subscale scores of walking, moderate and vigorous physical activity, and the score is categorized into "low", "medium", or "high" physical activity category.
MATRICS Consensus Cognitive Battery | 12 weeks (baseline and week 12)
  An evaluation of key cognitive domains relevant to individuals with schizophrenia
Investigation of Mental Rotation, Allocentricity-Egocentricity, and Perspective Taking (IMAP) | 12 weeks (baseline and week 12)
  An evaluation of the ability of participants to take perspective from an egocentric or allocentric point of view and to rotate mentally the stimulus or their point of view. Participants are rated on accuracy and reaction time.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Hahn, PhD, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre For Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hennekens CH, Hennekens AR, Hollar D, Casey DE. Schizophrenia and increased risks of cardiovascular disease. Am Heart J. 2005 Dec;150(6):1115-21. doi: 10.1016/j.ahj.2005.02.007. PMID 16338246
- [Background] Gold SM, Dziobek I, Sweat V, Tirsi A, Rogers K, Bruehl H, Tsui W, Richardson S, Javier E, Convit A. Hippocampal damage and memory impairments as possible early brain complications of type 2 diabetes. Diabetologia. 2007 Apr;50(4):711-9. doi: 10.1007/s00125-007-0602-7. Epub 2007 Feb 14. PMID 17334649
- [Background] Letourneau G, Bentaleb LA, Stip B, Luck D, Stip E. Relationships between Brain Structure and Metabolic Changes in Schizophrenia Patients Treated with Olanzapine: A Voxel-Based Morphometric Study. Schizophr Res Treatment. 2011;2011:862350. doi: 10.1155/2011/862350. Epub 2011 May 25. PMID 22937275
- [Background] Bora E, Akdede BB, Alptekin K. The relationship between cognitive impairment in schizophrenia and metabolic syndrome: a systematic review and meta-analysis. Psychol Med. 2017 Apr;47(6):1030-1040. doi: 10.1017/S0033291716003366. Epub 2016 Dec 29. PMID 28032535